CLINICAL TRIAL: NCT02611830
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study, With a Vedolizumab IV Reference Arm, to Evaluate the Efficacy and Safety of Vedolizumab Subcutaneous as Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis Who Achieved Clinical Response Following Open-Label Vedolizumab Intravenous Therapy
Brief Title: Efficacy and Safety of Vedolizumab Subcutaneously (SC) as Maintenance Therapy in Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002SC-3027; 2015-000480-14 (EudraCT Number); U1111-1168-0813 (Registry Identifier: WHO); 16/LO/0089 (Registry Identifier: NRES); NL55501.056.15 (Registry Identifier: CCMO); JapicCTI-163222 (Registry Identifier: JapicCTI); 189732 (Registry Identifier: HC-CTD); 163300410A0046 (Registry Identifier: NREC)
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Colitis, Ulcerative
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Maintenance Phase: Induction IV + Vedolizumab 108 mg SC (Experimental): Participants received vedolizumab 300 mg IV infusion in open-label induction phase and achieved clinical response at Week 6 were randomized to receive vedolizumab SC in maintenance phase. Vedolizumab SC, 108 mg, injection, Q2W and placebo-matching IV infusions, Q8W, starting at Week 6 up to approximately Week 50.
  Interventions: Drug: Vedolizumab 300 mg IV; Drug: Placebo IV; Drug: Vedolizumab 108 mg SC
- Maintenance Phase: Induction IV + Vedolizumab 300 mg IV (Experimental): Participants received vedolizumab 300 mg IV infusion in open-label induction phase and achieved clinical response at Week 6 were randomized to receive vedolizumab IV in maintenance phase. Vedolizumab 300 mg, IV infusion, Q8W and placebo-matching SC injection, Q2W starting at Week 6 up to approximately Week 50.
  Interventions: Drug: Vedolizumab 300 mg IV; Drug: Placebo SC
- Maintenance Phase: Induction IV + Placebo (Experimental): Participants received vedolizumab 300 mg IV infusion in open-label induction phase and achieved clinical response at Week 6 were randomized to receive placebo in maintenance phase. Placebo-matching subcutaneous (SC) injections, once every 2 weeks (Q2W) and placebo-matching IV infusions, once every 8 weeks (Q8W) starting at Week 6 up to approximately Week 50.
  Interventions: Drug: Vedolizumab 300 mg IV; Drug: Placebo IV; Drug: Placebo SC

INTERVENTIONS:
Drug: Vedolizumab 300 mg IV — Vedolizumab intravenous infusion
Drug: Placebo IV — Vedolizumab intravenous infusion placebo
  Arms: Maintenance Phase: Induction IV + Placebo; Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Drug: Vedolizumab 108 mg SC — Vedolizumab subcutaneous injection
  Arms: Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Drug: Placebo SC — Vedolizumab subcutaneous injection placebo
  Arms: Maintenance Phase: Induction IV + Placebo; Maintenance Phase: Induction IV + Vedolizumab 300 mg IV

SUMMARY:
The purpose of this study is to assess the effect of vedolizumab subcutaneous (vedolizumab SC) maintenance treatment on clinical remission at Week 52 in participants with moderately to severely active ulcerative colitis (UC) who achieved clinical response following administration of vedolizumab intravenous (vedolizumab IV) induction therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab subcutaneous (vedolizumab SC). Vedolizumab SC is being tested to treat people who have moderate to severely active ulcerative colitis. This study will look at clinical remission as well as mucosal healing, durable clinical response, durable clinical remission, and corticosteroid free remission in participants with UC who receive vedolizumab SC maintenance therapy after having achieved a clinical response to vedolizumab IV induction therapy.

The study enrolled 383 patients. All participants will enter into a 6-week Induction Phase where they will be administered open-label vedolizumab IV 300 mg via intravenous infusion (IV) at Week 0 (Day 1) and Week 2 (Day 15), and will then be assessed for a clinical response at Week 6. Participants who achieve a clinical response at Week 6 will be randomly assigned to one of the three treatment groups:

Vedolizumab SC 108 mg Q2W and Placebo IV Q8W Vedolizumab IV 300 mg Q8W and Placebo SC Q2W Placebo SC Q2W and Placebo IV Q8W

Participants who do not achieve a clinical response at Week 6 will not be randomized in to the Maintenance Period, and will receive a third infusion of vedolizumab IV 300 mg at Week 6.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 71 weeks (up to 4 weeks of screening, 52 weeks of treatment and 18 weeks of safety follow-up). Participants will make multiple visits to the clinic, plus a final visit 18 weeks after last dose of study drug for a follow-up assessment. Participants will also participate in a long-term safety follow-up, by phone, at 6 months after the last dose of study drug.

After the Week 52 assessments, participants meeting protocol-defined criteria were eligible to enroll in Study MLN0002SC-3030 (NCT02620046; Long-term Safety) to receive open-label vedolizumab treatment. Participants who withdrew early (prior to Week 52) due to sustained nonresponse, disease worsening, or the need for rescue medications may also have been eligible for Study MLN0002SC-3030. Participants who did not enroll into Study MLN0002SC-3030 were to complete a final on-study safety assessment at Week 68 (or final safety visit 18 weeks after the last dose) in the Maintenance Phase of Study MLN0002SC-3027.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ulcerative colitis (UC) established at least 6 months prior to screening, by clinical and endoscopic evidence and corroborated by a histopathology report.
2. Moderately to severely active UC as determined by a complete Mayo score of 6-12 (with an endoscopic subscore ≥2)
3. Evidence of UC extending proximal to the rectum (≥15 cm of involved colon).
4. Inadequate response with, loss of response to, or intolerance to corticosteroids, immunomodulators, or Tumor Necrosis Factor-alpha (TNF-α) antagonists

Exclusion Criteria:

1. Evidence of abdominal abscess or toxic megacolon at the initial Screening Visit.
2. Extensive colonic resection, subtotal or total colectomy.
3. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
4. Prior exposure to investigational or approved non-biologic therapies (eg, cyclosporine, tacrolimus, thalidomide, methotrexate or tofacitinib) for the treatment of underlying disease within 30 days or 5 half-lives of screening (whichever is longer).
5. Prior exposure to any investigational or approved biologic or biosimilar agent within 60 days or 5 half-lives of screening (whichever is longer).
6. Prior exposure to vedolizumab
7. Surgical intervention for UC required at any time during the study.
8. History or evidence of adenomatous colonic polyps that have not been removed or has a history or evidence of colonic mucosal dysplasia.
9. Suspected or confirmed diagnosis of Crohn's entercolitis, indeterminate colitis, ischaemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
10. Active infections
11. Chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection, HIV or tuberculosis (active or latent), identified congenital or acquired immunodeficiency. HBV immune participants (ie, being hepatitis B surface antigen [HBsAg] negative and hepatitis B antibody positive) may, however, be included.
12. History of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, demyelinating or neurodegenerative disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (174):
- United States (28):
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Rocky Mountain Clinical Research, LLC, Wheat Ridge, Colorado
  - Middlesex Gastroenterology Associates, Middletown, Connecticut
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - L & L Research Choices, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Research Concierge, LLC, Owensboro, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Metropolitan Gastroenterology Group, PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Long Island Clinical Research Associates, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Virginia Mason Seattle Main Clinic, Seattle, Washington
- Expertia S.A- Mautalen Salud e Investigacion, Ciudad Autonoma Buenos Aires, Argentina
- Australia (5):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (2):
  - Clinique Saint-Pierre, Ottignies
  - AZ Delta, Roeselare
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Brazil (4):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - HUCFF-UFRJ - Hospital Universitario Clementino Fraga Filho - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio Do Janeiro
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
- Bulgaria (8):
  - MHAT 'Avis Medica' OOD, Pleven
  - MHAT - Silistra AD, Silistra
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - Second MHAT - Sofia AD, Sofia
  - "City Clinic UMHAC" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Canada (3):
  - London Health Science Centre, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
- Czechia (5):
  - Ccbr-Synarc A/S, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - A-SHINE s.r.o., Pilsen
  - Ccbr-Synarc A/S, Prague
  - Axon Clinical, s.r.o., Prague
- Odense Universitetshospital, Odense C, Denmark
- West Tallinn Central Hospital, Tallinn, Estonia
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - EUGASTRO GmbH, Leipzig, Saxony
  - Krankenhaus Waldfriede e. V., Berlin
- Hungary (6):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (2):
  - Wolfson Medical Center, Holon
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (7):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (19):
  - Nagoya, Aichi-ken
  - Sakura-shi, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Nishinomiya-shi, Hyōgo
  - Takamatsu, Kagawa-ken
  - Kamakura-shi, Kanagawa
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Saga, Saga-ken
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Bunkyō City, Tokyo-To
  - Minatoku, Tokyo-To
  - Mitaka-shi, Tokyo-To
  - Shinjuku-ku, Tokyo-To
  - Wakayama, Wakayama
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Republican Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Mexico (6):
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - iBiomed Guadalajara, Zapopan, Jalisco
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Christus Muguerza Sur S.A. de C.V., Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Maastricht University Medical Center, Maastricht
- Poland (14):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - NZOZ Vitamed, Bydgoszcz
  - SP CSK im. prof. K. Gibinskiego SUM, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - SPZOZ Uniwersytecki Szpital Klin. nr 1 im.N.Barlickiego UM, Lodz
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - GASTROMED Sp. z o.o., Lublin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
- Romania (3):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Russia (9):
  - TSBIH "Territorial Clinical Hospital", Krasnoyarsk
  - FSBIH "Central Clinical Hospital of Russian Academy of Sciences", Moscow
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBI "Scientific Research Institute of Physyology and Basic Medicine" under the SB of RAMS, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - SBEI HPE "Rostov State Medical University" of the MoH of the RF, Rostov-on-Don
  - SPb SBIH "City Hospital of Saint Martyr Elizaveta", Saint Petersburg
  - LLC "RIAT SPb", Saint Petersburg
  - SBIH of Yaroslavl region " Regional Clinical Hospital ", Yaroslavl
- Serbia (5):
  - Clinical Center Zvezdara, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
- South Korea (5):
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
- Spain (2):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
- Sweden (2):
  - Karolinska Universitetssjukhuset - Solna, Stockholm
  - Danderyds Sjukhus AB, Stockholm
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty, Ankara
  - Acibadem Fulya Hospital, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
- Ukraine (13):
  - RCI Chernivtsi RCH Dep of Surgery Bukovinian SMU, Chernivtsi
  - SI Institute of Gastroenterology of NAMSU Dept of Stomach & Duodenum Diseases, D&ThN SI DMA of MoHU, Dnipro
  - Regional CH Dep of Gastroenterology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CHI Prof.O.O.Shalimov Kharkiv City Clinical Hospital #2, Kharkiv
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - CI A.and O. Tropiny City Clinical Hospital, Kherson
  - Kyiv CCH #12 Dept of Therapy O.O.Bogomolets NMU, Kyiv
  - MI of Healthcare Kyiv RCH P.L. Shupyk NMA of PGE, Kyiv
  - CI Odesa Regional Clinical Hospital, Odesa
  - SI Divisional Clinical Hospital of Uzhgorod Station of ST&BA LZ Dep of Therapy SHEI Uzhgorod NU, Uzhhorod
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - SI Branch CH of Zaporizhzhia Station-2 of SE Prydniprovska Railway Dept of Surgery Zaporizhzhia SMU, Zaporizhzhia
- United Kingdom (3):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Whipps Cross University Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] D'Haens G, Baert F, Danese S, Kobayashi T, Loftus EV Jr, Sandborn WJ, Dornic Q, Lindner D, Kisfalvi K, Marins EG, Vermeire S. Efficacy of vedolizumab during intravenous induction therapy in ulcerative colitis and Crohn's disease: post hoc analysis of patient-reported outcomes from the VISIBLE 1 and 2 studies. Eur J Gastroenterol Hepatol. 2024 Apr 1;36(4):404-415. doi: 10.1097/MEG.0000000000002728. Epub 2024 Feb 21. PMID 38417060
- [Derived] Kobayashi T, Ito H, Ashida T, Yokoyama T, Nagahori M, Inaba T, Shikamura M, Yamaguchi T, Hori T, Pinton P, Watanabe M, Hibi T. Efficacy and safety of a new vedolizumab subcutaneous formulation in Japanese patients with moderately to severely active ulcerative colitis. Intest Res. 2021 Oct;19(4):448-460. doi: 10.5217/ir.2020.00026. Epub 2020 Aug 18. PMID 32806876
- [Derived] Sandborn WJ, Baert F, Danese S, Krznaric Z, Kobayashi T, Yao X, Chen J, Rosario M, Bhatia S, Kisfalvi K, D'Haens G, Vermeire S. Efficacy and Safety of Vedolizumab Subcutaneous Formulation in a Randomized Trial of Patients With Ulcerative Colitis. Gastroenterology. 2020 Feb;158(3):562-572.e12. doi: 10.1053/j.gastro.2019.08.027. Epub 2019 Aug 28. PMID 31470005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one hundred forty-one investigative sites in North America, South America, Western/Northern Europe, Central Europe, Eastern Europe and Africa/Asia/Australia from 18-Dec-2015 to 21-Aug-2018.
Pre-assignment Details: A total of 383 participants were enrolled in open-label (OL) induction phase, 353 participants completed. 216 participants achieved clinical response at Week 6 were randomized into maintenance phase and participants who did not achieve clinical response at Week 6, received 3rd dose of open label vedolizumab IV 300 mg and completed Week 14 visit.
Groups:
- Open-Label Induction Phase: Vedolizumab 300 mg IV: Vedolizumab 300 mg, intravenous (IV) infusion, once at Weeks 0, 2 in the open-label induction phase.
Period: OL Induction Phase
Arm/Group | Open-Label Induction Phase: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Started | 383 | 0 | 0 | 0
Completed (Completers included randomized participants, or if not randomized, those who had Week 14 visit) | 353 | 0 | 0 | 0
Not Completed | 30 | 0 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 9 | 0 | 0 | 0
Not completed — Significant Protocol Deviation | 4 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 0 | 0 | 0
Not completed — Reason not specified | 3 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Open-Label Induction Phase: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Started (Participants who achieved clinical response at Week 6 entered the maintenance phase.) | 0 | 56 | 106 | 54
Completed | 0 | 20 | 75 | 39
Not Completed | 0 | 36 | 31 | 15
Not completed — Lack of Efficacy | 0 | 29 | 18 | 6
Not completed — Pretreatment Event/Adverse Event | 0 | 5 | 5 | 2
Not completed — Significant Protocol Deviation | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Voluntary Withdrawal | 0 | 1 | 2 | 5
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Reason not specified | 0 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of vedolizumab IV.
Groups:
- Vedolizumab IV 300 mg, Induction Phase Only: Vedolizumab 300 mg, intravenous (IV) infusion, once at Weeks 0, 2 in the open-label induction phase. Participants who did not achieve clinical response at Week 6 were not randomized into the maintenance phase and received a 3rd dose of vedolizumab 300 mg IV infusion at Week 6.
- Total: Total of all reporting groups
Arm/Group | Vedolizumab IV 300 mg, Induction Phase Only | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV | Total
Number analyzed (Participants) | 167 | 56 | 106 | 54 | 383
Age, Continuous [Mean (Full Range); unit: years] | 42.7 [18 to 79] | 39.4 [21 to 66] | 38.1 [18 to 69] | 41.6 [18 to 68] | 40.79 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 22 | 41 | 23 | 165
  Male | 88 | 34 | 65 | 31 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Non-Hispanic and Latino | 24 | 6 | 7 | 8 | 45
  Not Collected | 143 | 49 | 99 | 46 | 337
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
  Asian | 39 | 13 | 14 | 5 | 71
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 125 | 42 | 92 | 47 | 306
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 1 | 0 | 2 | 1 | 4
  Japan | 27 | 10 | 10 | 2 | 49
  Korea, Republic Of | 10 | 3 | 4 | 3 | 20
  Czech Republic | 2 | 3 | 10 | 4 | 19
  Hungary | 2 | 2 | 2 | 6 | 12
  Poland | 37 | 13 | 35 | 10 | 95
  Serbia | 1 | 1 | 0 | 1 | 3
  Slovakia | 3 | 0 | 4 | 3 | 10
  Bosnia | 0 | 0 | 2 | 0 | 2
  Bulgaria | 3 | 1 | 1 | 1 | 6
  Croatia | 8 | 1 | 0 | 1 | 10
  Estonia | 2 | 0 | 0 | 0 | 2
  Israel | 2 | 0 | 0 | 0 | 2
  Romania | 4 | 0 | 3 | 0 | 7
  Russia | 12 | 0 | 5 | 3 | 20
  Turkey | 1 | 2 | 0 | 0 | 3
  Ukraine | 11 | 4 | 6 | 2 | 23
  Canada | 4 | 3 | 2 | 2 | 11
  United States | 24 | 6 | 7 | 8 | 45
  Brazil | 4 | 0 | 3 | 1 | 8
  Mexico | 2 | 1 | 0 | 0 | 3
  Belgium | 0 | 2 | 0 | 0 | 2
  Denmark | 0 | 1 | 0 | 0 | 1
  Germany | 0 | 3 | 3 | 1 | 7
  Italy | 4 | 0 | 2 | 3 | 9
  Lithuania | 0 | 0 | 4 | 1 | 5
  Netherlands | 1 | 0 | 0 | 0 | 1
  Spain | 1 | 0 | 0 | 0 | 1
  United Kingdom | 1 | 0 | 1 | 1 | 3
Height [Mean (Full Range); unit: cm] | 169.3 [145 to 193] | 172.4 [147 to 194] | 171.9 [151 to 197] | 171.2 [152 to 196] | 170.7 [145 to 197]
Weight [Mean (Full Range); unit: kg] | 68.20 [37.0 to 150.2] | 73.96 [40.6 to 160.0] | 71.58 [44.0 to 131.0] | 76.95 [50.6 to 124.8] | 71.21 [37.0 to 160.0]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — Body Mass Index = weight/height
  kg/m^2 | 23.65 [15.1 to 40.3] | 24.66 [14.1 to 51.1] | 24.07 [17.0 to 41.0] | 26.21 [16.3 to 35.3] | 24.28 [14.1 to 51.1]
Female Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 17 | 4 | 3 | 8 | 32
  Surgically Sterile | 8 | 1 | 2 | 3 | 14
  Female of Childbearing Potential | 54 | 17 | 36 | 12 | 119
  Participant is a male | 88 | 34 | 65 | 31 | 218
Smoking Classification [Count of Participants; unit: Participants]
  Has never smoked | 107 | 38 | 70 | 33 | 248
  Is a current smoker | 7 | 0 | 11 | 10 | 28
  is an ex-smoker | 53 | 18 | 25 | 11 | 107
Duration of Ulcerative Colitis [Mean (Standard Deviation); unit: years] — Population: Data for duration of ulcerative colitis prior therapy was collected only for maintenance phase arm groups.
  years
    number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    (all) |  | 7.36 (7.147) | 7.96 (6.217) | 8.18 (5.929) | 7.86 (6.380)
Ulcerative Colitis Prior Therapy [Count of Participants; unit: Participants] — Population: Data for ulcerative colitis prior therapy was collected only for maintenance phase arm groups.
  Participants
    Without Prior Corticosteroids or Immunomodulators: number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Without Prior Corticosteroids or Immunomodulators: Yes |  | 1 | 1 | 0 | 2
    Without Prior Corticosteroids or Immunomodulators: No |  | 55 | 105 | 54 | 214
    Only Prior Corticosteroids: number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Only Prior Corticosteroids: Yes |  | 22 | 28 | 21 | 71
    Only Prior Corticosteroids: No |  | 34 | 78 | 33 | 145
    Only Prior Immunomodulators: number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Only Prior Immunomodulators: Yes |  | 1 | 6 | 1 | 8
    Only Prior Immunomodulators: No |  | 55 | 100 | 53 | 208
    With Prior Corticosteroids and Immunomodulators: number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    With Prior Corticosteroids and Immunomodulators: Yes |  | 32 | 71 | 32 | 135
    With Prior Corticosteroids and Immunomodulators: No |  | 24 | 35 | 22 | 81
Participants with Prior TNF-alpha Antagonist Use [Count of Participants; unit: Participants] — Population: Data for prior TNF-alpha antagonist use was collected only for maintenance phase arm groups.
  Participants
    number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Yes |  | 20 | 40 | 24 | 84
    No |  | 36 | 66 | 30 | 132
Participants with Prior TNF-alpha Antagonist Failure [Count of Participants; unit: Participants] — Population: Data for prior TNF-alpha antagonist failure was collected only for maintenance phase arm groups.
  Participants
    number analyzed (Participants) | 0 | 20 | 40 | 24 | 84
    (all) |  | 20 | 40 | 24 | 84
Participants with Prior Immunomodulator Failure and Prior TNF-alpha Antagonist Failure [Count of Participants; unit: Participants] — Population: Data for prior immunomodulator failure and prior TNF-alpha antagonist failure was collected only for maintenance phase arm groups.
  Participants
    number analyzed (Participants) | 0 | 17 | 34 | 19 | 70
    Yes |  | 12 | 21 | 13 | 46
    No |  | 5 | 13 | 6 | 24
Worst Prior Treatment Failure [Count of Participants; unit: Participants] — Anti-TNF failure includes all participants who failed an anti-TNF. Immunomodulator failure includes all participants who failed an immunomodulator but did not fail an anti-TNF. Corticosteroid failure includes all participants who failed a Corticosteroid and who did not fail an anti-TNF nor an Immunomodulator. Population: Data for worst prior treatment failure was collected only for maintenance phase arm groups.
  Participants
    Prior TNF-alpha Antagonist Failure: number analyzed (Participants) | 0 | 20 | 40 | 24 | 84
    Prior TNF-alpha Antagonist Failure: Inadequate Response |  | 9 | 21 | 13 | 43
    Prior TNF-alpha Antagonist Failure: Loss of Response |  | 8 | 17 | 9 | 34
    Prior TNF-alpha Antagonist Failure: Intolerance |  | 3 | 2 | 2 | 7
    Prior Immunomodulator Failure: number analyzed (Participants) | 0 | 5 | 22 | 5 | 32
    Prior Immunomodulator Failure: Inadequate Response |  | 1 | 6 | 2 | 9
    Prior Immunomodulator Failure: Loss of Response |  | 0 | 3 | 0 | 3
    Prior Immunomodulator Failure: Intolerance |  | 4 | 13 | 3 | 20
    Prior Corticosteroid Failure: number analyzed (Participants) | 0 | 13 | 23 | 15 | 51
    Prior Corticosteroid Failure: Inadequate Response |  | 5 | 14 | 5 | 24
    Prior Corticosteroid Failure: Loss of Response |  | 4 | 6 | 9 | 19
    Prior Corticosteroid Failure: Intolerance |  | 4 | 3 | 1 | 8
Baseline Disease Activity [Count of Participants; unit: Participants] — Population: Data for baseline disease activity was collected only for maintenance phase arm groups.
  Participants
    number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Moderate (Mayo Score=6 to 8) |  | 20 | 46 | 17 | 83
    Severe (Mayo Score=9 to 12) |  | 36 | 60 | 37 | 133
Baseline Fecal Calprotectin [Mean (Standard Deviation); unit: ug/g] — Population: Data for Baseline fecal calprotectin was collected only for maintenance phase arm groups. Number analyzed is the number of participants with data available for baseline fecal calprotectin.
  ug/g
    number analyzed (Participants) | 0 | 56 | 102 | 52 | 210
    (all) |  | 2393.4 (2859.66) | 2607.2 (2908.67) | 3173.5 (4785.48) | 2690.4 (3451.64)
Extraintestinal Manifestations [Count of Participants; unit: Participants] — Population: Data for extraintestinal manifestations was collected only for maintenance phase arm groups.
  Participants
    number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Yes |  | 5 | 13 | 7 | 25
    No |  | 51 | 93 | 47 | 191
Disease Localization [Count of Participants; unit: Participants] — Population: Data for disease localization was collected only for maintenance phase arm groups. Number analyzed is the number of participants with data available for disease localization.
  Participants
    number analyzed (Participants) | 0 | 56 | 105 | 54 | 215
    Proctosigmoiditis |  | 7 | 15 | 7 | 29
    Left Sided Colitis |  | 24 | 46 | 21 | 91
    Extensive Colitis |  | 4 | 7 | 7 | 18
    Pancolitis |  | 21 | 37 | 19 | 77
Corticosteroid Use at Baseline [Count of Participants; unit: Participants] — Population: Data for corticosteroid use at Baseline was collected only for maintenance phase arm groups. Number analyzed is the number of participants with data available for corticosteroid use at baseline.
  Participants
    number analyzed (Participants) | 0 | 56 | 106 | 54 | 216
    Yes |  | 24 | 45 | 21 | 90
    No |  | 32 | 61 | 33 | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 52
Description: Clinical remission is defined as a complete Mayo score ≤ 2 points and no individual subscore > 1 point. The Mayo score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 52
Population: The Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. Participants who only received induction IV therapy and were not randomized into the maintenance phase were not included in the FAS; participants were analyzed according to the randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Number analyzed (Participants) | 56 | 106 | 54
percentage of participants | 14.3 [6.4 to 26.2] | 46.2 [36.5 to 56.2] | 42.6 [29.2 to 56.8]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value was calculated by Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata according to concomitant use of corticosteroids, clinical remission status at Week 6, and previous TNF-α antagonist failure/concomitant immunomodulator; Risk Difference (RD) = 32.3, 95% CI 2-sided [19.7 to 45.0]

2. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 52
Description: Mucosal healing is defined as Mayo endoscopic subscore ≤1 point. The findings on endoscopy scale ranges from 0 to 3, where 0=normal or inactive disease 1=mild disease (erythema, decreased vascular pattern, mild friability) 2=moderate disease (marked erythema, lack of vascular pattern, friability, erosions) 3=severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 52
Population: The FAS included all randomized participants who received at least 1 dose of study drug. Participants who only received induction IV therapy and were not randomized into the maintenance phase were not included in the FAS; participants were analyzed according to the randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Number analyzed (Participants) | 56 | 106 | 54
percentage of participants | 21.4 [11.6 to 34.4] | 56.6 [46.6 to 66.2] | 53.7 [39.6 to 67.4]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value was calculated by CMH test stratified by randomization strata according to concomitant use of corticosteroids, clinical remission status at Week 6, and previous TNF-α antagonist failure/concomitant immunomodulator; Risk Difference (RD) = 35.7, 95% CI 2-sided [22.1 to 49.3]

3. Secondary Outcome: Percentage of Participants Achieving Durable Clinical Response at Week 6 and Week 52
Description: Durable clinical response is defined as clinical response at both Weeks 6 and 52, where clinical response is defined as a reduction in complete Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point. The Mayo score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Baseline, Weeks 6 and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Number analyzed (Participants) | 56 | 106 | 54
percentage of participants | 28.6 [17.3 to 42.2] | 64.2 [54.3 to 73.2] | 72.2 [58.4 to 83.5]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 36.1, 95% CI 2-sided [21.2 to 50.9]

4. Secondary Outcome: Percentage of Participants Achieving Durable Clinical Remission at Week 6 and Week 52
Description: Durable clinical remission is defined as clinical remission at both Weeks 6 and 52. Clinical remission is defined as a complete Mayo score of less than or equal to (≤) 2 points and no individual subscore greater than (>) 1 point. The Mayo score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Weeks 6 and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Number analyzed (Participants) | 56 | 106 | 54
percentage of participants | 5.4 [1.1 to 14.9] | 15.1 [8.9 to 23.4] | 16.7 [7.9 to 29.3]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; Test type: Superiority; p = 0.076, Fisher Exact — P-value was calculated by Fisher's Exact Test; Risk Difference (RD) = 9.7, 95% CI 2-sided [-6.6 to 25.7]

5. Secondary Outcome: Percentage of Participants Achieving Corticosteroid-free Remission at Week 52
Description: Corticosteroid-free remission is defined as participants using oral corticosteroids at Baseline (Week 0) who have discontinued oral corticosteroids and are in clinical remission at Week 52. Clinical remission is defined as a complete Mayo score of ≤ 2 points and no individual subscore > 1 point. The Mayo score is a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consists of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore is scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 52
Population: Participants from FAS, who used concomitant oral corticosteroid at Baseline. FAS included all randomized participants who received at least 1 dose of study drug and who only received induction IV therapy and were not randomized into maintenance phase were not included in FAS; participants were analyzed according to randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
Number analyzed (Participants) | 24 | 45 | 21
percentage of participants | 8.3 [1.0 to 27.0] | 28.9 [16.4 to 44.3] | 28.6 [11.3 to 52.2]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; Test type: Superiority; p = 0.067, Fisher Exact — P-value was calculated by Fisher's Exact Test; Risk Difference (RD) = 20.6, 95% CI 2-sided [-4.5 to 43.7]

ADVERSE EVENTS:
Time Frame: From first dose up to 18 weeks post last dose of study drug (Up to approximately 68 weeks)
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report AEs occurring at any other time during the study. Any adverse event reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vedolizumab IV 300 mg, Induction Phase Only | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/56 | 0/106 | 0/54
Serious Adverse Events (participants affected / at risk) | 17/167 | 6/56 | 10/106 | 7/54
Other Adverse Events (participants affected / at risk) | 34/167 | 31/56 | 42/106 | 31/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab IV 300 mg, Induction Phase Only (N=167) | Maintenance Phase: Induction IV + Placebo (N=56) | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC (N=106) | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV (N=54)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 12 | 5 | 3 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Drug resistance (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab IV 300 mg, Induction Phase Only (N=167) | Maintenance Phase: Induction IV + Placebo (N=56) | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC (N=106) | Maintenance Phase: Induction IV + Vedolizumab 300 mg IV (N=54)
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 5 | 5
Colitis ulcerative (Gastrointestinal disorders) | 7 | 14 | 12 | 5
Nasopharyngitis (Infections and infestations) | 4 | 11 | 11 | 10
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 10 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 2 | 0 | 4
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 6 | 4
Headache (Nervous system disorders) | 5 | 6 | 9 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT02611830/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02611830/SAP_000.pdf